CLINICAL TRIAL: NCT03335995
Title: Stroke Prognosis in Intensive CarE - The SPICE Registry
Brief Title: Stroke Prognosis in Intensive CarE
Acronym: SPICE
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C17-16
Record Dates: First submitted 2017-10-19; First posted 2017-11-08 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2021-08

CONDITIONS: Acute Stroke Patients Requiring Invasive Mechanical Ventilation
Keywords: mechanical invasive ventilation; course of the care; prognosis; stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The S.P.I.C.E registry is an investigator-initiated prospective multicenter cohort study which will be conducted in 35 ICUS in the Paris area.The aim of the study is to determine the trajectory of acute stroke patients requiring invasive mechanical ventilation, focusing on functional outcomes at 3 months and 1 year following ICU admission. This project is funded by the French Agence Régionale de Santé (ARS).

ELIGIBILITY:
Inclusion criteria:

* Age>18 years
* Acute stroke (acute ischaemic stroke, brain hemorrhage, subarachnoid hemorrhage). The stroke diagnosis date is defined by the date of the initial brain imaging (TDM or MRI).
* Admitted to ICU within 7 days before or after the diagnosis of stroke.
* Requiring invasive mechanical ventilation in ICU for more than 24 hours.

Exclusion criteria:

* Traumatic causes of stroke
* Refusal of the patient, or his reliable person, to participate in the study.
* Privation of liberty by administrative or judicial decision

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects included in this study are adult patients requiring invasive mechanical ventilation at the acute phase of stroke (within 7 days of stroke onset), irrespective of indication for intubation.
  Prolonged mechanical ventilation of several days to weeks in ICU may be required for some patients, with various ICU discharge trajectories in survivors.
Sampling Method: Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2020-11-18 (Actual)

PRIMARY OUTCOMES:
Functional outcome | One year
  Score on the modified Rankin scale (a disability score that ranges from 0 [no symptoms] to 6 [death]). Patients will be classified as "good outcome" (score of 0-3) or poor outcome (score of 4-6, indicating severe disability or death).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François TIMSIT, Study Director — U 1137
Locations (1):
- Bichat Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sonneville R, Mazighi M, Collet M, Gayat E, Degos V, Duranteau J, Gregoire C, Sharshar T, Naim G, Cortier D, Jost PH, Foucrier A, Bagate F, de Montmollin E, Papin G, Magalhaes E, Guidet B, Ben Hadj Salem O, Benghanem S, le Guennec L, Delpierre E, Legriel S, Megarbane B, Toumert K, Tran M, Geri G, Monchi M, Bodiguel E, Mariotte E, Demoule A, Zarka J, Diehl JL, Roux D, Barre E, Tanaka S, Osman D, Pasquier P, Lamara F, Crassard I, Boursin P, Ruckly S, Staiquly Q, Timsit JF, Woimant F; SPICE Investigators. One-Year Outcomes in Patients With Acute Stroke Requiring Mechanical Ventilation. Stroke. 2023 Sep;54(9):2328-2337. doi: 10.1161/STROKEAHA.123.042910. Epub 2023 Jul 27. PMID 37497675
- [Background] Sonneville R, Mazighi M, Bresson D, Crassard I, Crozier S, de Montmollin E, Degos V, Faugeras F, Gayat E, Josse L, Lamy C, Magalhaes E, Maldjian A, Ruckly S, Servan J, Vassel P, Vigue B, Timsit JF, Woimant F; SPICE investigators. Outcomes of Acute Stroke Patients Requiring Mechanical Ventilation: Study Protocol for the SPICE Multicenter Prospective Observational Study. Neurocrit Care. 2020 Apr;32(2):624-629. doi: 10.1007/s12028-019-00907-0. PMID 32026446